CLINICAL TRIAL: NCT05591456
Title: Accelerated Hypofractionated 1 Week Radiotherapy in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rawda Ahmed Abdul Hakim Balata, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Radiotherapy in Breast Cancer
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer Radiotherapy
MeSH Terms: interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: The patients who met the inclusion criteria were randomly divided into two groups, each group of 50 patients. The first group (arm A) will receive a dose of 27 Gy to the chest wall using 3D conformal radiotherapy (5.4 Gy per fraction) over one week, whilst, the second group (arm B) will receive a dose of 40 Gy to the chest wall (2.67 Gy per fraction) over three weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): The first group 50 patient (arm A) will receive a dose of 27 Gy to the chest wall using 3D conformal radiotherapy (5.4 Gy per fraction) over one week,
  Interventions: Radiation: adjuvant radiotherapy
- group 2 (Active Comparator): the second group 50 patient (arm B) will receive a dose of 40 Gy to the chest wall (2.67 Gy per fraction) over three weeks.
  Interventions: Radiation: adjuvant radiotherapy

INTERVENTIONS:
Radiation: adjuvant radiotherapy — Treatment schedule and delivery The patients who met the inclusion criteria were randomly divided into two groups, each group of 50 patients. The first group (arm A) will receive a dose of 27 Gy to the chest wall using 3D conformal radiotherapy (5.4 Gy per fraction) over one week, whilst, the second group (arm B) will receive a dose of 40 Gy to the chest wall (2.67 Gy per fraction) over three weeks.

SUMMARY:
Accelerated hypofractionated 1 week post-mastectomy chest wall irradiation in breast cancer patients will presumably produce comparable toxicity and disease control in comparison to 3 weeks schedule.

The aim is to evaluate toxicity and disease control after implementation of accelerated hypofractionated 1 week chest wall irradiation in breast cancer patients.

DETAILED DESCRIPTION:
Operational Design Patient Assessment Pre-radiotherapy assessment is done to provide a baseline for use in further follow-up and to rule out metastasis. This includes detailed history taking, full physical examination, hematological and biochemical laboratory evaluation, tumor markers: CA15-3, plain chest X-ray, pelvi-abdominal ultrasound, ECHO for left cancer breast, bone scan if indicated.

Treatment schedule and delivery The patients who met the inclusion criteria were randomly divided into two groups, each group of 50 patients. The first group (arm A) will receive a dose of 27 Gy to the chest wall using 3D conformal radiotherapy (5.4 Gy per fraction) over one week, whilst, the second group (arm B) will receive a dose of 40 Gy to the chest wall (2.67 Gy per fraction) over three weeks.

Setup, simulation and target definition For setup, patients were positioned on a wingboard with both arms raised above the head and radiopaque markers along breast borders. Subsequently, the 5-mm slice-thick axial CT images were acquired from the lower mandible aspect to 5 cm below contralateral inframammary fold. The CT images will be automatically transferred to a planning workstation, where the CTV and relevant organs-at-risk (OARs) will be outlined. The planning of the tangential fields will be based on the target volume delineation for the dose-volume distribution analysis. The heart and ipsilateral lung were separately contoured as organs at risk, the heart was outlined to the pulmonary trunk superiorly, including pericardium and excluding major vessels. For setup verification purposes, weekly digitally reconstructed radiographs (DRRs) were performed.

Evaluation of Treatment Follow-up is done for assessment of toxicity and disease-free and overall survival.

During follow-up, patients are examined after completion of radiotherapy and at 3 and 6 months. Surveillance includes a full clinical examination, hematological and biochemical laboratory evaluation, tumor markers: CA15-3, plain chest X-ray, pelvi-abdominal ultrasound, ECHO for left cancer breast, bone scan if indicated.

Acute skin toxicity was assessed at the completion of radiotherapy and after 3 months (RTOG 2015), late skin toxicity was scored from 6 months after radiation and referred to the time of last examination (LENT/Soma Tables 1995). The maximal detected toxicity was scored according to the Common Terminology Criteria for Adverse Events, version 3.0, using the RTOG/EORTC toxicity scale associated with radiation as reference (NCI 2013) (Cox et al, 1995).

Admininistrative Design

Approvals for performing this study are obtained from:

A) The recruited cases; B) The Institutional Review Board (IRB) RESULTS Collected data will be presented in tables and suitable graphs and analyzed using SSPS package. Mean and standard deviations will be estimated for quantitative data and median for non-normally distributed data. Actuarial or life tables analysis will be used for estimating survival and long-rank test for comparison of curves. P value is significant at 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of breast adenocarcinoma
* prior modified radical mastectomy
* negative resection margins (3 mm)
* pathological stage pT1-pT2, N0-2 (AJCC, 2017)
* no macroscopic evidence of distant metastases at diagnosis
* Age 18-80 years
* Normal hematological and biochemical laboratory tests
* Written informed consent was obtained from all patients

Exclusion Criteria:

* locally advanced disease pT3-pT4, N3
* positive surgical margins
* prior thoracic radiation
* synchronous second primary tumor
* distant metastases
* pregnancy
* presence of a concomitant psychiatric disorder precluding an aware informed consent.
* age >80 years

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
detection of breast shrinkage | three months after radiotherapy
  breast size measured before and after radiotharapy
detection of breast shrinkage | 6 months after radiotherapy
  breast size measured before and after radiotharapy
breast on the treated side is indurated | 3 months after radiotherapy
  the induration detected by palpation with comparison with the normal side
detection of irregularity of breast shape | 3 months after radiotherapy
  change in the normal shape of the breast detected by inspection and photogaphing before and after radiotherapy
breast on the treated side is indurated | 6 months after radiotherapy
  the induration detected by palpation with comparison with the normal side
detection of irregularity of breast shape | 6 months after radiotherapy
  change in the normal shape of the breast detected by inspection and photogaphing before and after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Balata, dr, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ash DV, Benson EA, Sainsbury JR, Round C, Head C. Seven-year follow-up on 334 patients treated by breast conserving surgery and short course radical postoperative radiotherapy: a report of the Yorkshire Breast Cancer Group. Clin Oncol (R Coll Radiol). 1995;7(2):93-6. doi: 10.1016/s0936-6555(05)80808-8. PMID 7619770
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Fajdic J, Djurovic D, Gotovac N, Hrgovic Z. Criteria and procedures for breast conserving surgery. Acta Inform Med. 2013 Mar;21(1):16-9. doi: 10.5455/AIM.2013.21.16-19. PMID 23572855
- [Background] Aleknavicius E, Atkocius V, Kuzmickiene I, Steponaviciene R. Postmastectomy internal mammary nodal irradiation: a long-term outcome. Medicina (Kaunas). 2014;50(4):230-6. doi: 10.1016/j.medici.2014.09.010. Epub 2014 Oct 7. PMID 25458960
- [Background] Mannino M, Yarnold JR. Shorter fractionation schedules in breast cancer radiotherapy: clinical and economic implications. Eur J Cancer. 2009 Mar;45(5):730-1. doi: 10.1016/j.ejca.2009.01.024. Epub 2009 Feb 23. No abstract available. PMID 19243933